CLINICAL TRIAL: NCT05742737
Title: Frailty Index as An Indicator Associated With Postoperative Adverse Outcomes In The Older Population
Status: Completed | Type: Observational
Sponsor: Weidong Mi (Other)
Responsible Party: Sponsor-Investigator, Weidong Mi, Director of anesthesiology department, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: PLAGH-Frailty
Record Dates: First submitted 2023-01-27; First posted 2023-02-24 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robust: Unlike previous frailty index, mFI-5 uses a small number of variables readily available in a patient's history, including functional status (partial or complete dependence), history of diabetes, COPD, congestive heart failure, and hypertension requiring medication. 1 point is assigned to each variable. Functional status refers to needing some or all of the assistance of others in daily activities, including bathing, eating, dressing, going to the toilet, moving, traveling, and more. The mFI-5 score was calculated by increasing the number of variables per patient Patients were divided into 3 groups based on their mFI-5: frail group (mFI-5, 2-5) , prefrail group (mFI-5, 1) and robust group (mFI-5, 0). The range of the mFI-5 is from 0 to 5 with increments of 1, and increasing the mFI-5 implies increasing frailty.
- Prefrail: Unlike previous frailty index, mFI-5 uses a small number of variables readily available in a patient's history, including functional status (partial or complete dependence), history of diabetes, COPD, congestive heart failure, and hypertension requiring medication. 1 point is assigned to each variable. Functional status refers to needing some or all of the assistance of others in daily activities, including bathing, eating, dressing, going to the toilet, moving, traveling, and more. The mFI-5 score was calculated by increasing the number of variables per patient Patients were divided into 3 groups based on their mFI-5: frail group (mFI-5, 2-5) , prefrail group (mFI-5, 1) and robust group (mFI-5, 0). The range of the mFI-5 is from 0 to 5 with increments of 1, and increasing the mFI-5 implies increasing frailty.
  Interventions: Other: Frailty Index
- frail: Unlike previous frailty index, mFI-5 uses a small number of variables readily available in a patient's history, including functional status (partial or complete dependence), history of diabetes, COPD, congestive heart failure, and hypertension requiring medication. 1 point is assigned to each variable. Functional status refers to needing some or all of the assistance of others in daily activities, including bathing, eating, dressing, going to the toilet, moving, traveling, and more. The mFI-5 score was calculated by increasing the number of variables per patient Patients were divided into 3 groups based on their mFI-5: frail group (mFI-5, 2-5) , prefrail group (mFI-5, 1) and robust group (mFI-5, 0). The range of the mFI-5 is from 0 to 5 with increments of 1, and increasing the mFI-5 implies increasing frailty.
  Interventions: Other: Frailty Index

INTERVENTIONS:
Other: Frailty Index — The mFI-5 scoring system used in the current study was developed by Saxton and Velanovich by comparing the five variables in the original CSHA-FI with NSQIP database
  Groups: Prefrail; frail

SUMMARY:
This study is a observational study in China, which aims to explore the predictive effect of preoperative frailty defined by the modified frailty index in predicting postoperative survival and complications in elderly patients.

The objectives of the study include:

1. To demonstrate that the frailty scale can predict short- and long-term survival after surgery in elderly surgical patients; 2 Demonstrated that frailty as defined by this scale is associated with postoperative complications in older patients

DETAILED DESCRIPTION:
Traditionally, frailty has been described as the form of chronological age. Evaluating the patient's risks based solely on age is difficult, several other factors contribute to physiologic aging and determine functional reserve and response to the risk of postoperative complications. To meet the clinical demand for simpler frailty measurement tools, a simplified 5-index modified frailty index (mFI-5) has been proposed and validated in many literatures. However, there is a lack of evidence on the link between preoperative weakness and poor prognosis in elderly patients undergoing non cardiac surgery.

Therefore, the purpose of this study is to verify the prognostic value of mFI-5 for short-term and long-term adverse outcomes such as postoperative delirium, anxiety, depression, acute pain, and mortality in elderly non-cardiac surgery patients. Our hypothesis is that frailty may be highly correlated with postoperative mortality and adverse outcomes in elderly patients undergoing non-cardiac surgery, and that mFI-5 may be an effective risk prediction tool for decision-making and surgical planning.

ELIGIBILITY:
Inclusion Criteria:

(1) participants ≥ 65 years of age;

Exclusion Criteria:

1. lacked any covariate indicator or missing data for any confounder (such as demographic information, intraoperative surgery or anesthesia information);
2. ASA physical status Ⅴ;
3. Anesthesia other than general intravenous anesthesia or intravenous inhalation anesthesia;
4. Surgery time ≤ 60 min.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The lack of sufficient study data, however, does not demonstrate a dose-response relationship, with higher frailty levels having a greater impact on mortality [9]. Accordingly, this article would focus on the relationship between patients with varying degrees of frailty and long-term postoperative adverse outcomes and how preoperative planning and interventions can alter surgical trajectories and associated outcomes. According to our hypothesis, preoperative frailty can provide prognostic information, in addition to frequently recognized risks and consequences.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
12-month all-cause mortality | postoperative 12-month
  12-month postoperative mortality in elderly patients over 65 years of age
6-month all-cause mortality | postoperative 6-month
  6-month postoperative mortality in elderly patients over 65 years of age
1-month all-cause mortality | postoperative 1-month
  1-month postoperative mortality in elderly patients over 65 years of age

SECONDARY OUTCOMES:
Readmission rates | postoperative 30-day
  The rate of second admissions in elderly patients over 65 years old who underwent surgery within 30 days after surgery
Admission to ICU | From the moment of living operation room to the moment of discharge from hospital,up to 7 day
  Elderly surgical patients over the age of 65 are admitted to the intensive care unit after surgery
major complications | From the moment of living operation room to the moment of discharge from hospital,up to 7 day
  Postoperative complications include delirium, anxiety, depression, acute pain, stroke, major adverse cardiac events, acute kidney injury, infection, etc

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No